CLINICAL TRIAL: NCT00004254
Title: Phase II Study on Tomusex in Malignant Mesothelioma
Brief Title: Raltitrexed in Treating Patients With Malignant Mesothelioma That Cannot Be Surgically Removed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-08992; EORTC-08992
Record Dates: First submitted 2000-01-28; First posted 2004-04-23 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — raltitrexed

INTERVENTIONS:
Drug: raltitrexed

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of raltitrexed in treating patients who have malignant mesothelioma that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the therapeutic activity and toxicities of raltitrexed in patients with inoperable malignant mesothelioma. II. Determine the objective response rate and duration of response in patients treated with this regimen.

OUTLINE: This is a multicenter study. Within 2 weeks of staging procedures, patients receive raltitrexed IV over 15 minutes on day 1. Treatment repeats every 3 weeks for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks until disease progression and then every 8 weeks thereafter for survival.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven inoperable malignant mesothelioma All tumor stages eligible At least 1 target lesion with measurable disease in at least 1 dimension (20 cm or more with conventional techniques OR 10 cm or more with spiral CT scans) Outside irradiated field Prior surgery allowed if evidence of disease progression thereafter No signs or symptoms of CNS metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ZUBROD/ECOG/WHO 0-2 (after palliative measures such as pleural drainage) Life expectancy: Not specified Hematopoietic: Hemoglobin at least 10.0 g/dL WBC at least 4,000/mm3 Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.46 mg/dL Albumin at least 3.0 g/dL ALT and AST less than 2.5 times upper limit of normal (ULN) (less than 5 times ULN if liver involvement) Renal: Creatinine less than 1.69 mg/dL Creatinine clearance at least 65 mL/min Other: No other malignancies (including melanoma, hypernephroma, or breast carcinoma) within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception No uncontrolled infection No psychologic, familial, sociologic, or geographic condition that could interfere with compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent anticancer immunotherapy before first disease progression Chemotherapy: No prior systemic or intracavitary cytotoxic drugs No concurrent intrapleural or other systemic cytotoxic drugs Endocrine therapy: No concurrent anticancer hormonal agents (except corticosteroids) before first disease progression Radiotherapy: See Disease Characteristics Concurrent palliative radiotherapy allowed for painful lesions, needle tracts, or surgical scars or prevention of metastases along biopsy tracks At least 4 weeks since prior radiotherapy No prior radiotherapy to sole indicator lesion unless lesion is clearly progressive Surgery: See Disease Characteristics Prior pleurodesis allowed except with cytotoxic drugs (e.g., bleomycin) Concurrent pleurodesis with noncytotoxic drugs allowed Other: At least 1 month since other prior investigational agent No other concurrent anticancer agents before first disease progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-11; Primary Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD, PhD, Study Chair — Free University Medical Center
Locations (6):
- Italy (4):
  - Ospedale Bellaria, Bologna
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Universita Degli Studi di Udine, Udine
- Netherlands (2):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam

REFERENCES:
- [Background] Francart J, Legrand C, Sylvester R, Van Glabbeke M, van Meerbeeck JP, Robert A. Progression-free survival rate as primary end point for phase II cancer clinical trials: application to mesothelioma--The EORTC Lung Cancer Group. J Clin Oncol. 2006 Jul 1;24(19):3007-12. doi: 10.1200/JCO.2005.05.1359. PMID 16809726
- [Result] Baas P, Ardizzoni A, Grossi F, Nackaerts K, Numico G, Van Marck E, van de Vijver M, Monetti F, Smid-Geirnaerdt MJ, van Zandwijk N, Debruyne C, Legrand C, Giaccone G; EORTC Lung Cancer Group. The activity of raltitrexed (Tomudex) in malignant pleural mesothelioma: an EORTC phase II study (08992). Eur J Cancer. 2003 Feb;39(3):353-7. doi: 10.1016/s0959-8049(02)00668-8. PMID 12565988